CLINICAL TRIAL: NCT04276909
Title: Feasibility of the LUM Imaging System for Detection of Primary Pancreatic Cancer and Peritoneal Invasion From Primary Pancreatic Cancer During Surgery
Brief Title: Feasibility Study of LUM Imaging System for Pancreatic Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not initiated.
Sponsor: Lumicell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLP-00011
Record Dates: First submitted 2019-08-12; First posted 2020-02-19 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Pancreatic Cancer
Keywords: Primary Pancreatic Cancer; Peritoneal Invasion
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Lum Imaging System (Experimental): Single dose of LUM015 (1.0 mg/kg) will be administered by intravenous injection at the beginning of the surgery. All subjects will have intraoperative imaging using the LUM Imaging Device
  Interventions: Combination Product: LUM Imaging System

INTERVENTIONS:
Combination Product: LUM Imaging System — LUM015 will be administered at the beginning of surgery. All subjects will have intraoperative imaging using the LUM imaging device.

SUMMARY:
This single-site, non-randomized, open-label study to assess the initial safety and efficacy of the LUM Imaging System for detection of primary pancreatic cancer and peritoneal invasion from primary pancreatic cancer during surgery. In this feasibility study, the tumor detection algorithm will be developed for this indication.

DETAILED DESCRIPTION:
This study is being conducted to see if LUM015 can be safely given to human patients before surgery at a dose that allows the removed tumor tissue to be identified when imaged by the LUM imaging device.

Up to 30 subjects will be enrolled in this study. Subjects will be administered with LUM015 at a dose of 1.0 mg/kg. Due to the expected duration of these surgeries (up to 14 hours), all subjects will require LUM015 administration intraoperatively.

The sequence of events during the surgical procedure will vary based on the standard of care used by the surgeon. Study treatment ends when the surgery is completed. All patients will continue their enrollment in the study until their first follow-up visit and they will continue to be followed until the medical team determines no further surgical intervention is required. Patients with adverse events that are determined to be possibly related to the LUM Imaging System will be followed until resolution or stabilization of the adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histological or cytological confirmation of pancreatic cancer on a biopsy prior to the operation with planned surgical resection. Subjects at any cancer stage will be enrolled.
* Age of 18 years or older.
* Subjects must be able and willing to follow study procedures and instructions.
* Subjects must have received and signed an informed consent form.
* Subjects must be otherwise healthy except for the diagnosis of cancer, as per the exclusion criteria listed below.
* Subjects must have normal organ and marrow function as defined below:
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 100,000/mcL
* AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels above institutional normal.
* Subjects with ECOG performance status of 0 or 1.

Exclusion Criteria:

* Subjects who are pregnant or nursing at the time of diagnosis
* Subjects who are sexually active and not willing/able to use medically acceptable forms of contraception (hormonal or barrier method of birth control, abstinence) upon entering the study and for 60 days after injection of LUM015.
* Subjects who have taken an investigational drug within 30 days of enrollment.
* Subjects who have not recovered from adverse events due to other pharmaceutical or diagnostic agents.
* Subjects with uncontrolled hypertension defined as persistent systolic blood pressure > 180 mm Hg, or diastolic blood pressure > 100 mm Hg; those subjects with known HTN should be under these values while under pharmaceutical therapy.
* History of allergic reaction attributed to drugs containing polyethylene glycol (PEG).
* History of allergic reaction to any oral or intravenous contrast agents.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, COPD or asthma requiring hospitalization within the past 12 months, or psychiatric illness/social situations that would limit compliance with study requirements.
* Subjects with QT interval > 470 ms.
* HIV-positive individuals on combination antiretroviral therapy are ineligible.
* Any subject for whom the investigator feels participation is not in the best interest of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Assess the initial safety and efficacy of the LUM Imaging System for detection of primary pancreatic cancer and peritoneal invasion from primary pancreatic cancer during surgery | 10-14 days
  Reported adverse events will be assessed and aggregated according to event type, relation to device or drug, and severity.

SECONDARY OUTCOMES:
Correlate resected tissue with LUM Imaging System to identify imaging threshold | 10-14 days
  Findings from imaging results with the LUM System will be correlated with pathology assessment of the resected tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ferrone, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No